CLINICAL TRIAL: NCT05768893
Title: Evaluation of Combined Treatment With Er:YAG Laser and Long-pulsed Nd:YAG Laser for the Treatment of Recalcitrant Warts: a Prospective Randomized Controlled Trial
Brief Title: Evaluation of Combined Treatment With Er:YAG & Nd:YAG Lasers for the Treatment of Recalcitrant Warts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0141-21-RMB
Record Dates: First submitted 2023-02-26; First posted 2023-03-15 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Viral Wart
Keywords: viral warts; recalcitrant; treatment; Er:YAG laser; long-pulsed Nd:YAG laser
MeSH Terms: conditions — Warts | interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial included 240 lesions from 24 patients diagnosed with recalcitrant warts. Each wart of the 240 was given a number and photographed. In cases when the patient had an uneven number of warts, one wart was excluded randomly. Then, the warts of each patient were randomly divided into two groups using computerized randomization and assigned to group 1 or group 2. Each group consisted of 120 warts.
  Group 1: Combined Er:YAG laser and long-pulsed Nd:YAG laser group. Group 2: Er:YAG laser group.
Who Masked: Outcomes Assessor
Masking Description: The primary assessor was given two photographs of each lesion, the first is the unmarked photograph copy (doesn't indicate to what group each lesion belongs) that was taken prior to the procedure, the second is the photograph that was taken in the follow up 5 weeks later. Assessments based on the two photographs were conducted by the primary assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1: Combined Er:YAG laser and long-pulsed Nd:YAG laser group (Experimental): This group included 120 wart lesions, treated with Er:YAG laser followed by LP Nd:YAG laser after 1-2 minutes. Cryo 6 (Zimmer Medizin Systems) was used to cool the lesions before, during and after applying the Nd:YAG laser.
  Interventions: Device: Long-Pulsed Nd:YAG Laser 1064nm & Er:YAG Laser 2940nm
- Group 2: Er:YAG laser group. (Active Comparator): This group included 120 wart lesions, treated with Er:YAG laser only.
  Interventions: Device: Er:YAG Laser 2940nm

INTERVENTIONS:
Device: Long-Pulsed Nd:YAG Laser 1064nm & Er:YAG Laser 2940nm — Warts with this intervention treated firstly with the Er:YAG laser, followed by the Nd:YAG laser in the same session.
  Arms: Group 1: Combined Er:YAG laser and long-pulsed Nd:YAG laser group
Device: Er:YAG Laser 2940nm — Warts with this intervention treated only with the Er:YAG laser.
  Arms: Group 2: Er:YAG laser group.

SUMMARY:
Background: Viral warts are common infectious skin disease induced by human papillomavirus (HPV). Lasers have been used for warts treatment in recent years with variable success rates.

Objective: The goal of this clinical trial is to prospectively evaluate combined treatment with Er:YAG laser and long-pulsed Nd:YAG laser compared to Er:YAG laser for the treatment of recalcitrant warts after one session. The main question it aims to answer is:

Does adding a treatment of long-pulsed Nd:YAG laser to Er:YAG laser in the same treatment session to the same wart have more curing effect than using the Er:YAG laser alone? This study included 240 lesions from 24 patients. All the lesions were diagnosed clinically as recalcitrant warts after failure of topical treatment and Cryotherapy. 120 lesions underwent a combined therapy of Er:YAG and long-pulsed (LP) Nd:YAG lasers, and the remaining 120 lesions underwent Er:YAG laser therapy only. The clearance rate was evaluated 5 weeks after and classified by three-graded evaluation: complete response, partial response, and poor response.

Researchers will compare the 120 treated warts with the combined lasers therapy to the 120 treated warts treated with Er:YAG laser alone to see if adding the Nd:YAG laser therapy has an additional curing value.

DETAILED DESCRIPTION:
Viral warts are benign epithelial proliferations, characteristically 1-20 mm in diameter, that develop secondary to infection of keratinocytes by human papilloma virus (HPV). HPV comprises a large group of approximately 120 genotypes that infect the epithelia of the skin or mucosa. Warts are a common dermatological complaint, with an estimated incidence of 5%-20% in children and adults, with peak incidence reported during teenage years. Patients often express a significant reduction in quality of life due to this cosmetic nuisance, as well as functional problems and physical discomfort when they occur on the palms of the hands and soles of the feet. Therefore, cutaneous warts are one of the most common pathologies treated by the clinical dermatologist.

Although warts may eventually spontaneously disappear once the immune system ﬁnds a way to eradicate the virus, the time taken for this to occur varies and can range from months to years. Managing recalcitrant warts may require more than one treating session. Chemical destruction can be induced with salicylic acid, cantharidin, formaldehyde, or glutaraldehyde, among other agents. Chemotherapeutic agents include podophyllin, podophyllotoxin, 5-fluorouracil, and bleomycin. Allergic contact agents used against recalcitrant warts include dinitrochlorobenzene and squaric acid dibutyl ester. More recently, immunomodulators such as interferon, systemic retinoids, cimetidine, and topical imiquimod have been used. The used methods of physical destruction include surgical excision, electrodesiccation, cryosurgery, and pulsed dye or carbon dioxide laser therapy.

Most of the methods mentioned above have their drawbacks and side effects. Surgical methods have proven somewhat effective but have their disadvantages of pain and long recovery periods and may offer incomplete and superficial results leading to high recurrence rates. Topical management requires the application of drugs for long durations and treatment success is, therefore, highly dependent on patient compliance.

Lasers are new methods of energy-based devices for treating warts. Er:YAG laser (like CO2 laser) is an ablative laser emitting at a wavelength of 2940 nm and highly absorbed by water. It is considered a safe treatment for viral warts, However, in many patients, mainly those with plantar warts, a significant rate of relapse may occur, requiring additional therapy. Recently, the long-pulsed (LP) 1064 nm Nd:YAG laser has attracted attention in the treatment of palmoplantar warts. The mechanism of the LP Nd:YAG laser is different from the Er:YAG laser. It targets the dermal blood vessels that supply infected cells and destroy them via photothermolysis mechanism. However, the limitations of this method are that the treatment usually requires several sessions, and the clearance rate after one session ranges between 14-22%.

This prospective study evaluates the treatment efficacy of an Er:YAG laser alone compared to a combination of Er:YAG followed by LP Nd:YAG after one session of recalcitrant warts. The investigators hypothesize that combining the two mechanisms of ablating the wart and coagulating the blood supply may lead to a higher wart clearance rate after a sole treatment session.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were clinically diagnosed with recalcitrant warts after two or more failed treatment lines with Cryotherapy and topical treatments.
2. Patients above the age of 8 and under the age of 80.

Exclusion Criteria:

1. The use of topical treatment for wart lesions in the past month.
2. Methods of physical destruction of the lesions in the past month such as surgical excision, electrodesiccation, cryosurgery or laser were excluded.
3. Patients with single wart lesion were excluded.
4. Pregnant and breast- feeding patients.
5. Patients on anticoagulant drugs.
6. Children below the age of 8.

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Comparison of the curing rate of the treatment between the two groups. | 5 weeks following the treatment.
  The cure rate of the treatment was classified by a three-grade evaluation according to the clearance at the end of therapy:
  * Complete response was considered when 100% of the wart disappeared.
  * Partial response was considered when 50-99% of the wart was disappeared.
  * Poor response was considered when less than 50% of the wart was disappeared.
  The disappeared portion of the wart was estimated visually based on two photographs, the first taken minutes before the treatment, and second taken 5 weeks after the treatment.

SECONDARY OUTCOMES:
Side effects | 5 weeks following the treatment.
  Including Blisters, Crusts, Escars, Hypopigmentation, Hyperpigmentation, Hypertrophic scars.
Age of the patient. | 5 weeks following the treatment.
  Assess any correlations between the curing rate and age of the patient. This will be tested with a generalized linear model, namely a random intercept logistic regression that accounts for patient differences.
Gender of the patient. | 5 weeks following the treatment.
  Assess any correlations between the curing rate and gender of the patient. This will be tested with a generalized linear model, namely a random intercept logistic regression that accounts for patient differences.
Location of the warts. | 5 weeks following the treatment.
  Assess if there is any correlations between the curing rate location of the wart. the warts locations that were tested: Palmar, Plantar, Periungual.
  This will be tested with a generalized linear model, namely a random intercept logistic regression that accounts for patient differences.

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Khamaisi, MD, Study Director — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
Risk of re-identification of participant data, reuse of data for purposes that had not been approved by patients, or for unfair commercial purposes.

REFERENCES:
- [Background] Iranmanesh B, Khalili M, Zartab H, Amiri R, Aflatoonian M. Laser therapy in cutaneous and genital warts: A review article. Dermatol Ther. 2021 Jan;34(1):e14671. doi: 10.1111/dth.14671. Epub 2020 Dec 29. PMID 33314577
- [Background] Zorman A, Koron N. Wart removal without anesthesia using long-pulse 1064-nm Nd:YAG laser. J Cosmet Dermatol. 2021 Feb;20(2):506-512. doi: 10.1111/jocd.13593. Epub 2020 Jul 16. PMID 32640061
- [Background] Azizjalali M, Ghaffarpour G, Mousavifard B. CO(2) Laser therapy versus cryotherapy in treatment of genital warts; a Randomized Controlled Trial (RCT). Iran J Microbiol. 2012 Dec;4(4):187-90. PMID 23205250
- [Background] El-Mohamady Ael-S, Mearag I, El-Khalawany M, Elshahed A, Shokeir H, Mahmoud A. Pulsed dye laser versus Nd:YAG laser in the treatment of plantar warts: a comparative study. Lasers Med Sci. 2014 May;29(3):1111-6. doi: 10.1007/s10103-013-1479-y. Epub 2013 Nov 12. PMID 24218179
- [Background] Cobb MW. Human papillomavirus infection. J Am Acad Dermatol. 1990 Apr;22(4):547-66. doi: 10.1016/0190-9622(90)70073-q. PMID 2156916
- [Background] Hsu VM, Aldahan AS, Tsatalis JP, Perper M, Nouri K. Efficacy of Nd:YAG laser therapy for the treatment of verrucae: a literature review. Lasers Med Sci. 2017 Jul;32(5):1207-1211. doi: 10.1007/s10103-017-2219-5. Epub 2017 May 2. PMID 28466193
- [Background] El-Tonsy MH, Anbar TE, El-Domyati M, Barakat M. Density of viral particles in pre and post Nd: YAG laser hyperthermia therapy and cryotherapy in plantar warts. Int J Dermatol. 1999 May;38(5):393-8. doi: 10.1046/j.1365-4362.1999.00719.x. PMID 10369554
- [Background] Oni G, Mahaffey PJ. Treatment of recalcitrant warts with the carbon dioxide laser using an excision technique. J Cosmet Laser Ther. 2011 Oct;13(5):231-6. doi: 10.3109/14764172.2011.606465. PMID 21774662
- [Background] Brodell RT, Bredle DL. The treatment of palmar and plantar warts using natural alpha interferon and a needleless injector. Dermatol Surg. 1995 Mar;21(3):213-8. doi: 10.1111/j.1524-4725.1995.tb00155.x. PMID 7712088
- [Background] Yilmaz E, Alpsoy E, Basaran E. Cimetidine therapy for warts: a placebo-controlled, double-blind study. J Am Acad Dermatol. 1996 Jun;34(6):1005-7. doi: 10.1016/s0190-9622(96)90279-0. PMID 8647965